CLINICAL TRIAL: NCT07215208
Title: Abutment Health and Occlusal Analysis of CAD-CAM and Conventional Metallic Partial Denture Framework in Mandibular Kenedy Class III Cases: A Randomized Cross Over Clinical Trial
Brief Title: Abutment Analysis of Metallic Denture Frameworks in Mandibular Kenedy Class III Cases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samah Ahmed Abdallah Sharaka, PhD degree student, Prosthetic Dentistry Department, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Abutment analysis CAD-CAM
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: Occlusion; Prosthesis Durability
MeSH Terms: conditions — Bites and Stings; Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: - Prospective, randomized controlled, two-phase, crossover trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Operators, participants, and statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM metallic partial denture frameworks (Experimental): The digital technology makes it much easier in fabricating the prosthesis, so by the aid of this technology we can make accurate occlusal scan and jaw relation without annoying of the patient with the impression material. The software makes it much easier in designing and planning for proper established removable metallic partial denture, with one tap we can print the designed wax pattern and continue in the conventional steps of manufacturing the metallic partial denture
  Interventions: Other: CAD/CAM metallic partial denture frameworks
- Conventional metallic partial denture frameworks (Active Comparator): The conventional fabricated metallic partial dentures have been the standard method for fabricating the metallic frameworks. It is a reliable treatment option for the partially edentulous patients and the most commonly used for it is advantageous. The advantages of conventional metallic partial dentures are it considered to be more rigid even if in thin sections, has higher stiffness and strength, thanks to good thermal conductivity of metal it can conduct heat and cold, can be designed to minimize tissue coverage
  Interventions: Other: Conventional metallic partial denture frameworks

INTERVENTIONS:
Other: CAD/CAM metallic partial denture frameworks — The CAD/CAM workflow starts with scanning of the physical model (master cast) to create a 3D virtual representation. Dental professionals then digitally analyze this virtual model and design the metallic partial denture frameworks using specialized computer software. Once the design is finalized, a wax pattern of the framework is either milled or 3D printed. Then proceeding with this wax pattern to fabricate the final metal partial denture framework, either by conventional casting process, or milling of the metallic framework
  Arms: CAD/CAM metallic partial denture frameworks
Other: Conventional metallic partial denture frameworks — The metallic partial denture frameworks have proven to be affordable and convenient treatment option for partially dentate patients for it is rigidity and durability. It can be used in thin sections and provide high strength and stiffness. However, metallic partial denture frameworks also come with several drawbacks. A significant concern for some patients is the metallic display, which can lead to poor esthetics. Other disadvantages include increased prosthesis weight, a potential metallic taste, and a tendency for plaque accumulation. Additionally, they can induce stresses on the abutment teeth
  Arms: Conventional metallic partial denture frameworks

SUMMARY:
This study is aimed to compare CAD/CAM (digitally fabricated) metallic partial denture frameworks to conventionally fabricated metallic partial denture frameworks in mandibular Kennedy class-III arches in terms of abutment health and occlusal analysis

DETAILED DESCRIPTION:
Traditional metallic partial dentures with cobalt-chromium frameworks and clasps considered a reliable choice because they're affordable, durable and have a resistance to distortion. However, the fabrication of traditional metallic partial dentures involves several manual steps, like pouring of the stone casts, surveying the hard tissue and soft tissue undercuts to choose the best path of insertion, and meticulously waxing each component (major and minor connectors, rests, clasps, and denture base retainers) directly onto the cast. This hands-on process can result in some fabrication errors, which by in turn can increase the stresses on the teeth supporting the denture (abutments) and even other non-abutment teeth.

CAD/CAM technology is increasingly being used for the fabrication of metallic partial denture frameworks; it has been highlighting in several investigations. The workflow starts with an intra oral digital scan of the oral cavity, to generate a 3D digital model, that allows for electronic surveying. The metallic partial denture frameworks are then designed virtually using specialized software, after which a wax pattern is created by milling or rapid prototyping. Then the wax pattern would be casted conventionally into metallic partial denture frameworks. The key advantages are simplifying the fabrication process, enhance the accuracy of fit, and reduce the stresses on abutment teeth, significant time savings, and reduction of the potential errors inherent in traditional multi-step lab procedures

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral bounded saddles in the mandible (Kennedy class III).
* Opposing dentition is fully intact or restored.
* Sufficient inter-arch space.
* Angle's class I maxilla-mandibular relationship.

Exclusion Criteria:

* Periodontal affection of the abutment teeth.
* Skeletal mal-relation.
* Unmotivated patients to maintain adequate oral hygiene to follow up.
* Patients with neuromuscular and Psychiatric disorders.
* Systematic disease affecting bone and periodontal health.
* Insufficient inter-arch space.
* Patients with physical disabilities that could affect follow up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Abutment health mobility | 3 months
  Periotest, Periotest value (PTV) which ranges from -8 to +50

SECONDARY OUTCOMES:
Gingival bleeding index | 3 months
  Löe and Silness Gingival Index (GI), GI scale (scores) 0 -3 (with 0 being normal and 3 being severe inflammation)

OTHER OUTCOMES:
Occlusal Analysis | 3 months
  OccluSense Device, Force distribution per tooth